CLINICAL TRIAL: NCT01157130
Title: Prescriptive Exercise Intervention During Active Treatment for Early Stage Breast Cancer Patients: A Breast Cancer Rehabilitation & Exercise Laboratory
Brief Title: Breast Cancer Patients: A Breast Cancer Rehabilitation and Exercise Laboratory
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nevada Cancer Institute (Other)
Collaborators: Vons (Unknown)
Responsible Party: Karen Milligan, MD, Nevada Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NVCI 10-09
Record Dates: First submitted 2010-07-01; First posted 2010-07-05 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Early Stage Breast Cancer (Stage 0-III)
Keywords: Breast Cancer; Exercise; CRP; C-reactive protein; BMI; Nevada Cancer Institute; Rehabilitation; Prescriptive exercise; Physical Activity; DEXA; Obesity; lifestyle intervention; Early Stage Breast Cancer Patients (stage 0-III)
MeSH Terms: conditions — Breast Neoplasms; Motor Activity; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (Experimental): Each patient will have a weekly goal of 2000 calories burned and 18 MET-hours of exercise which can be achieved in 4 to 7 hours of physical activity per week. Resistance training, using weight machines and aerobic training using treadmills, elliptical trainers and stationary bicycles, will be utilized in the intervention group.
  Interventions: Other: Exercise Regimen
- Control Group (No Intervention): The control group will receive basic information on physical activity but not be instructed.

INTERVENTIONS:
Other: Exercise Regimen — Exercise instruction
  Arms: Intervention Group

SUMMARY:
The proposed study compares the outcomes of a physical activity intervention begun at diagnosis, continuing through active cancer treatment and into six months of survivorship compared to the outcomes of a control group receiving limited information on activity.

DETAILED DESCRIPTION:
Patients (with stage 0 to stage III breast cancer)receiving chemotherapy, radiation or both chemotherapy and radiation will be included in the study.Randomization will be stratified by disease stage at diagnosis, treatment modalities planned, and hormonal status. Each patient will have a weekly goal of 2000 calories burned and 18 MET-hours of exercise which can be achieved in 4 to 7 hours of physical activity per week. Resistance training, using weight machines and aerobic training using treadmills, elliptical trainers and stationary bicycles, will be utilized in the intervention group. The control group will receive basic information on physical activity but not be instructed. Any physical activity in this group will be self-reported. Change in C-reactive protein will be the primary endpoint. Changes in other laboratory values, DEXA measurements, and quality of life measurements will be secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Consent to participate in study
2. Women aged 18 and older
3. Stage 0 to III breast cancer prior to any treatment and at time of diagnosis
4. Requires treatment that includes chemotherapy, radiation therapy or both chemotherapy and radiation therapy
5. Adequate fitness to participate in a physical activity as assessed by the investigator
6. Willing and able to participate in a prescribed exercise program

Exclusion Criteria:

1. Metastatic breast cancer (Stage IV)
2. Initiation of treatment regimen prior to enrollment
3. Treatment for breast cancer not requiring chemotherapy or radiation therapy
4. Patients who are pregnant (negative urine pregnancy test required at baseline to determine eligibility in women of child bearing potential).
5. Currently lactating
6. Do not read, understand, or speak English

Eligible participants will not be included if they have:

1. known cardiac disease,
2. uncontrolled hypertension,
3. uncontrolled thyroid disease,
4. diabetes mellitus,
5. mental illness,
6. infection,
7. immune or endocrine abnormality,
8. body weight reduction I10% in past 6 months, and
9. positive exercise stress test.
10. Major surgery within last 6 months that requires exercise restriction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-07

PRIMARY OUTCOMES:
Changes in CRP
  The primary endpoint for this study change in C-reactive protein.

SECONDARY OUTCOMES:
Change in laboratory values
  Compare changes in:
  * Glucose
  * Insulin
  * Estradiol
  * Testosterone
Change in body composition
  Body composition parameters and bone density will be assessed using Dual Energy X-ray Absorptiometry (DEXA) and compared between the two groups.
Quality of Life
  Quality of Life will be measured and compared between the groups
Overall Survival
  Comparing overall survival and progression free survival between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Milligan, MD, Principal Investigator — Nevada Cancer Institute
Locations (1):
- Nevada Cancer Institute, Las Vegas, Nevada, United States

REFERENCES:
- See also: Nevada Cancer Institute — http://www.nevadacancerinstitute.org/